CLINICAL TRIAL: NCT05566106
Title: Anal Follow-up of Patients With a Gynecological History of High-grade Lesion and More Induced HPV
Acronym: Cohorte_HPV
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Cohorte_HPV
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Human Papilloma Virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human Papillomavirus (HPV) infection is the most common sexually transmitted infection in the world. It is currently estimated that 4.5% of all cancers worldwide are attributable to HPV, representing 630,000 new cases per year. HPV is responsible for more than 98% of pre-cancerous and cancerous lesions of the cervix and vagina and 88% of anal cancers.

Although prevention of HPV infection has been available since 2007, there are approximately 3000 new cases of cervical cancer in France each year. Women benefit from organized screening for cervical cancer.

HPV is also responsible for anal cancer in more than 90% of cases, mostly caused by HPV 16/18. Its incidence is lower with 1162 cases in women in 2018 but is increasing strongly (+88% in women since 1990).

As with cervical cancer, there are precursors to anal cancer: high-grade intraepithelial lesions. Early diagnosis of these lesions could potentially reduce the incidence of anal cancer, but there are still few data in the literature. The prevalence of anal carriage in patients with a history of cervical dysplasia or cervical cancer is estimated in studies to be 20% with a risk of high grade anal lesions of 8%.

The relative risk of developing anal cancer in women with a history of high-grade cervical lesions is about 5 per 100,000, 15 per 100,000 for those with a history of cervical cancer, and 42 and 48 per 100,000 respectively for women with HPV-induced pre-cancer and cancerous lesions of the vulva.

The different means of cervico-vaginal screening: screening samples: HPV test, cytology, some biomarkers: double labelling p16/ki67, E6-E7 mRNA and clinical examination with or without colposcopy (examination of the cervix with a magnifying glass) are used at the gynecological level but also at the anal level with as examination: simple anuscopy and high resolution anuscopy. Some scientific societies have established surveillance algorithms for certain risk groups, but there are no clinical practice recommendations yet for women with a history of gynecological HPV-induced lesions.

A proctology follow-up protocol for at-risk patients is proposed to patients based on cervico-vaginal surveillance recommendations and data in the literature, pending clinical practice guidelines. The frequency of these examinations depends on the patient's age and the existence of other risk factors for the development of anal HPV lesions. Depending on these elements, follow-up is proposed every 3 years, 5 years, or annually.

The objective of this work is therefore to propose proctological surveillance to this population considered at risk, according to age, smear results and HPV test.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with a high-grade or higher HPV-induced gynecological lesion
* Patient participating in the proctology follow-up protocol
* French-speaking patient

Exclusion Criteria:

* Patient with a history of induced high-grade anal HPV lesion and above
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient whose age ≥ 18 years, with a high-grade or higher HPV-induced gynecological lesion and participating in the proctology follow-up protocol.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2032-08-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of developing HPV-induced lesions | Year1
  This outcome corresponds to the number of HPV-induced lesions detected at the anal level according to the proctological follow-up protocol.

SECONDARY OUTCOMES:
Model for screening and anal follow-up in patients with a history of gynecologic high-grade HPV-induced lesions | Year 1
  This outcome corresponds to the comparison of time to onset of anal HPV-induced lesions in the study population at follow-up during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Wylomanski, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Clifford GM, Georges D, Shiels MS, Engels EA, Albuquerque A, Poynten IM, de Pokomandy A, Easson AM, Stier EA. A meta-analysis of anal cancer incidence by risk group: Toward a unified anal cancer risk scale. Int J Cancer. 2021 Jan 1;148(1):38-47. doi: 10.1002/ijc.33185. Epub 2020 Jul 29. PMID 32621759
- [Background] Islami F, Ferlay J, Lortet-Tieulent J, Bray F, Jemal A. International trends in anal cancer incidence rates. Int J Epidemiol. 2017 Jun 1;46(3):924-938. doi: 10.1093/ije/dyw276. PMID 27789668
- [Background] Abramowitz L, Lacau Saint Guily J, Moyal-Barracco M, Bergeron C, Borne H, Dahlab A, Bresse X, Uhart M, Cancalon C, Catella L, Benard S. Epidemiological and economic burden of potentially HPV-related cancers in France. PLoS One. 2018 Sep 20;13(9):e0202564. doi: 10.1371/journal.pone.0202564. eCollection 2018. PMID 30235216
- [Background] de Martel C, Plummer M, Vignat J, Franceschi S. Worldwide burden of cancer attributable to HPV by site, country and HPV type. Int J Cancer. 2017 Aug 15;141(4):664-670. doi: 10.1002/ijc.30716. Epub 2017 Jun 8. PMID 28369882